CLINICAL TRIAL: NCT03507946
Title: Single Center, Randomized, Blinded, Controlled Trial Evaluating the Safety and Effectiveness of Combined 460nm, 633nm and 830nm LED Light for the Treatment of Mild to Moderate Plaque-Type Psoriasis Vulgaris
Brief Title: Safety and Effectiveness of Combined LED Light for the Treatment of Mild to Moderate Plaque Type Psoriasis Vulgaris
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and sponsor decided to not pursue clinical trial
Sponsor: Ismart (Industry)
Responsible Party: Principal Investigator, Steven Baker, Principle Investigator, Ismart
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: version 2.1 March 24th 2018
Record Dates: First submitted 2018-04-09; First posted 2018-04-25 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Intervention Model Description: Randomized, Blinded, Controlled Trial
Masking Description: Randomization will be conducted by the study coordinator and will take place in a separate room away from the PI.
  The Study coordinator will number the 2 plaques 1 and 2. The Study coordinator will draw a sequential envelope containing the randomization code for the control and test. The code will inform the study coordinator which plaque is control and which test.
  The Study coordinator will complete the randomization coding worksheet which identifies the test and control plaque and location.
  The randomization coding worksheet will be kept separate from the subjects' case report form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test (Experimental): Subject self control; Plaque 1: Dermawrap - combined 460nm, 633nm, and 830nm LED therapyDaily treatments of 15 minutes of combined LED phototherapy, 5 days per week for 12 weeks.
  Plaque 2: No Intervention
  Interventions: Device: Dermawrap - combined 460nm, 633nm and 830nm LED therapy

INTERVENTIONS:
Device: Dermawrap - combined 460nm, 633nm and 830nm LED therapy — Daily treatments of 15 minutes of combined LED phototherapy, 5 days per week for 12 weeks.

SUMMARY:
The purpose of this study is to investigate whether light therapy can help improve plaque psoriasis. This is a study based on a new medical device. The device produces its light from light emitting diodes. This type of technology has been used for several years in the treatment of other skin conditions. However, the investigators want to study the effect of a combination of very specific wavelengths of light on reducing the signs and symptoms of plaque psoriasis.

The Investigators are looking to recruit 25 volunteers from the general population between the ages of 18 and 65 years old with mild to moderate plaque psoriasis and who are otherwise healthy. The light treatments are 5 times a week for 12 weeks and the treatment is self-administered at home. Each treatment is 15 minutes. The total duration of the study is 16 weeks.

This is a controlled trial. This means that the volunteer will treat one plaque with the light therapy device and the other plaque will remain untreated for the period of the study.

DETAILED DESCRIPTION:
This is a single center, randomized, blinded, interindividual, study involving 25 healthy subjects. After informed consent, confidentiality and photographic release forms, volunteers who meet all inclusion criteria and none of the exclusion criteria on page 4, will be entered into the study. Subjects with a PASI of ≤10 will be included in the study.

At Baseline, the Principle Investigator will identify comparable study plaques (where possible the plaques should be of comparable size, duration and severity and where possible on comparable body areas).

The plaques will be evaluated using the Localised Psoriasis Severity Index (LPSI).

At this point and thereafter, the Principle Investigator will be blinded to the intervention/plaque.

The plaques will be numbered 1 and 2 by the study coordinator. The plaques will then be randomised by the study coordinator to receive either the active treatment or act as the control.

Subjects test and control plaque will undergo a mechanical evaluation of hyperpigmentation and erythema using a MC1000® (Courage and Khazaka).

Subjects will complete a Dermatology Life Quality Index (DLQI) based on their psoriasis.

After randomization subjects will be instructed on how to use the Dermawrap device and the treatment schedule (5 x weekly treatments for 12 weeks).

A topical emollient (Hydrogel) will be dispensed to the subject and the subject will be instructed on its use and frequency (2 x weekly treatments for 12 weeks).

The Subjects were then be asked to carry out a self-treatment in front of the study staff. Subjects will be instructed on potential side effects and severity and encouraged to contact the research center in relation to any side effects or concerns.

Subjects will be given a subject diary to complete daily to capture any adverse incidents and record their treatment and treatment experiences.

Seven (7) (+/- 7days) after Baseline, subjects will be contacted by study staff to check for any adverse incidents or problems in using the device. Subjects will be asked if there has been any change in their health or medication from their last visit.

Twenty-eight (28) days (+/- 7days) after Baseline subjects will return to the study center. Subjects will be asked if there has been any change in their health or medication from their last visit. The PI will be notified of any changes. Any changes will be evaluated by the PI or SC against the exclusion criteria and recorded. Subjects diary will be collected and reviewed by the study staff for any adverse incidents.

Subjects test and control plaque will undergo a mechanical evaluation of hyperpigmentation and erythema using a MC1000® (Courage and Khazaka). Subjects test and control plaque will be photographed.

The device will be checked, and usage data will be collected from the device. The topical emollient (Hydrogel) will be dispensed to the subject.

Fifty-six (56) days (+/- 7days) after baseline subjects return to the study center for assessment. Subjects will be asked if there has been any change in their health or medication from their last visit. The PI will be notified of any changes. Any changes will be evaluated by the PI or SC against the exclusion criteria and recorded. Subjects diary will be collected and reviewed by the study staff for any adverse incidents The device will be checked, and usage data will be collected from the device. Subjects test and control plaque will be evaluated using the Localised Psoriasis Severity Index (LPSI) by the Blinded PI and will undergo a mechanical evaluation of hyperpigmentation and erythema using a MC1000® (Courage and Khazaka).

Subjects test and control plaque will be photographed Subjects will complete a Dermatology Life Quality Index (DLQI) based on their psoriasis. The topical emollient (Hydrogel) will be dispensed to the subject.

Eighty-four (84) days (+/- 7days) after baseline subjects return to the study center for assessment. Subjects will be asked if there has been any change in their health or medication from their last visit. The PI will be notified of any changes. Any changes will be evaluated by the PI or SC against the exclusion criteria and recorded.

Subjects diary will be collected and reviewed by the study staff for any adverse incidents The device will be collected from the subject, will be checked, and usage data will be collected from the device. The device will not be returned to the subject.

Subjects test and control plaque will be evaluated using the Localised Psoriasis Severity Index (LPSI) by the Blinded PI and will undergo a mechanical evaluation of hyperpigmentation and erythema using a MC1000® (Courage and Khazaka).

Subjects test and control plaque will be photographed Subjects will complete a Dermatology Life Quality Index (DLQI) based on their psoriasis. In addition, the subject will be asked to complete a standardized system usability scale (SUS). At day 84 (+/- 7 days) the subject will stop treatment.

One hundred and twelve (112) days (+/- 7days) the subject will return to the study center. Subjects will be asked by the Research assistant or Study coordinator if they have experienced any changes in their health or taken new/adjusted current medications since the last visit. The PI will be notified of any changes. Any changes will be evaluated by the PI or SC against the exclusion criteria and recorded. Subjects diary will be collected and reviewed by the study staff for any adverse incidents.

Blinded physician (PI) assessment of psoriasis plaques using the Localised Psoriasis Severity Index (LPSI), mechanical evaluation of hyperpigmentation and erythema using MC1000® (Courage and Khazaka).

Standardised digital photography and Subject self-assessment of treatment response Including Dermatology Life Quality Index (DLQI) will be conducted. Unless any AE or SAE have been reported and ongoing the subject will be signed out of the study.

The duration of subject participation is 16 weeks. The total duration of the study is expected to be 12 months to include recruitment of subjects.

ELIGIBILITY:
Inclusion Criteria:

Healthy male & females; 18 to 65 years of age with mild to moderate psoriasis ≤10 PASI according to the Psoriasis Area Severity Index.

Plaques comparable in terms of size, duration and severity and where possible on comparable body areas according to the localized psoriasis severity index (LPSI).

Fitzpatrick, I-V photo type skin types. Written informed consent is given. Volunteers agree NOT to use any over the counter or prescriptive psoriasis treatments during the study period unless specifically advised by the research staff.

Exclusion Criteria:

Volunteers who suffer from Erythrodermic, exfoliative or pustular psoriasis. Volunteers who suffer from a systemic photosensitive disorder such as Lupus erythematosus, photosensitive eczema or Albinism.

Volunteers who suffer from genetic deficiencies that increase susceptibility to dermatologic cancer such as Xeroderma pigmentosum.

Volunteers who suffer from diffuse actinic damage of the skin. Volunteers who suffer from localised fungal or bacterial skin infections in or around the treatment area.

Volunteers currently taking (or a history of taking) medication listed in Photosensitive drug list in instructions for use.

Subjects who have any known allergies to the ingredients in the emollient used in the study.

Volunteers with known malignancy and or undergoing chemotherapy, radiotherapy or high doses of corticosteroids.

Volunteer suffers from keloid scars, or birthmarks in the treatment area. Females who are pregnant, breastfeeding or who wish to become pregnant during the study period.

Enrolled in another clinical trial during the same study period. The volunteer has a planned hospital admission and/or surgical procedure for an illness or disease which existed before enrolment into the clinical trial and which may interfere with the course or outcome of the study.

The volunteer has a medical or psychological condition(s) associated with a risk of poor protocol compliance (e.g. alcoholism or drug abuse).

A volunteer is undergoing or is likely to undergo other treatments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of the local psoriasis severity index (LPSI) compared to the control area at the end of treatment | 84 days from baseline
  A change from baseline of the local psoriasis severity index (LPSI) compared to the control area at the end of treatment period (84 days)

SECONDARY OUTCOMES:
Change from baseline of the local psoriasis severity index (LPSI) compared to the control area at the end of study period | 112 days from baseline
  A change from baseline of the local psoriasis severity index (LPSI) compared to the control area 28 days after the end of the treatment.

OTHER OUTCOMES:
Safety evaluation; number of adverse incidents, evaluation of pigmentation of skin. | Baseline onwards
  Number of adverse incidents including reporting on hyperpigmentation of skin.

IPD SHARING:
Plan to Share IPD: No